CLINICAL TRIAL: NCT04285697
Title: The Impact of An Infection Prevention Bundle on Surgical Site Infections in Brain Tumor Surgery
Brief Title: Infection Prevention Bundle in Brain Tumor Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic, elevtive sugeries were temproraily delayed in our country. It's targeted to take cases again as of August 2020
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Fatma Balci, principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulUC
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Surgical Site Infection; Brain Tumor
Keywords: Care Bundles,; Surgical Wound Infection,; craniyal surgery; nursing care
MeSH Terms: conditions — Surgical Wound Infection; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Experimental): During the outpatient clinic visit, an information leaflet will be given about the subjects that should be considered for prevention of SSI before surgery. 2% mupirocin ointment will be applied to the nostrils with the swab twice-daily before surgery and once on the morning of surgery. Body cleaning will be done with 4% chlorhexidine gluconate shower the night before the surgery. Prophylactic antibiotics by weight will be administered within 60 minutes of anesthesia induction. The planned aseptic technique will be applied and a strict draping will be used in the incision site. Body temperature, blood pressure, respiratory rate, heart rate and O2 saturation of the patients will be monitored every 1 hour during the operation and data will be recorded on the data collection form. Before the skin closes, the surgical site will be washed with warm Isotonic NaCl solution. Wound care education will be provided to the patient and family before discharge.
  Interventions: Other: infection prevention bundle
- group 2 control (No Intervention): The pre-operative service sociodemographic characteristics form, preoperative, intra and postoperative evaluation forms will be completed. Body temperature, blood pressure, respiratory rate, heart rate and O2 saturation of the patients will be monitored every 1 hour during the operation and data will be recorded on the data collection form.

INTERVENTIONS:
Other: infection prevention bundle — The infection prevention bundle (IPB) implemented items:
  Preoperative counseling and questionnaire: patient counseling and preparation instructions, screening questions for signs of infection, and presence of open or nonhealing wounds.
  Nasal methicillin-resistant and methicillin-sensitive Staphylococcus aureus decolonization: preoperative 24 hours ago twice-daily application of 2% mupirocin ointment to bilateral nares with final application on the morning of surgery.
  Body decolonization: Cleansing with 4% chlorhexidine gluconate shower the evening before surgery and the morning of surgery.
  Preoperative weight-based antibiotics within 60 minutes of incision
  Strict draping and surgical techniques the standardization Irrigation of the surgical site with warm Isotonic NaCl solution before skin closure Postoperative wound care education to patient and family
  Arms: group 1

SUMMARY:
This study aimed to evaluate the effectiveness of an infection prevention bundle on surgical site infections in patients undergone brain tumor surgery. The patients were divided into 2 groups: infection prevention bundle group and control group

DETAILED DESCRIPTION:
In cranial neurosurgery, surgical site infections (SSIs) occur in 0.5%-7.2% of patients, frequently require reoperations and long-lasting antibiotic treatment, and are often life threatening.

Patients with malignant brain tumors often harbor several potential risk factors for SSI such as advanced age, poor nutritional state owing to appetite loss, poor sanitary condition of the head skin due to low performance status, immunosuppression caused by steroid or chemotherapeutic agents, and surgical site skin problems caused by post-operative irradiation. Therefore, patients with malignant brain tumors theoretically are a high-risk group for SSI.

A care bundle technique, which is an aggregate of evidence-based practices expected to improve patient outcomes, has been introduced to reduce the incidence of SSI.

The infection prevention bundle (IPB) implemented items:

1. Preoperative counseling and questionnaire: patient counseling and preparation instructions, screening questions for signs of infection, and presence of open or nonhealing wounds.
2. Nasal methicillin-resistant and methicillin-sensitive Staphylococcus aureus decolonization: preoperative 24 hours ago twice-daily application of 2% mupirocin ointment to bilateral nares with final application on the morning of surgery.
3. Body decolonization: Cleansing with 4% chlorhexidine gluconate shower the evening before surgery and the morning of surgery.
4. Preoperative weight-based antibiotics within 60 minutes of incision
5. Strict draping and surgical techniques the standardization
6. Irrigation of the surgical site with warm Isotonic NaCl solution before skin closure
7. Postoperative wound care education to patient and family

Care bundle in preventing surgical site infections is an approach that requires team-based service delivery and physician-nurse cooperation. Although it is known abroad and use of existing care bundle is not a new concept in Turkey, much is unknown, it is determined that widespread and effective use. Experimental studies on the care bundles are needed especially in our country to prevent surgical site infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists score I-II-III
* Surgical intervention planned with the diagnosis of brain tumor
* No systemic infection such as sepsis, pneumonia, blood infections, or intracranial infection such as meningitis, abscess or local infection.
* Not having a mental illness

Exclusion Criteria:

* Being morbidly obese (BMI> 40kg / m2)
* Immune deficiency
* Using immunosuppressive drugs
* Being addicted to alcohol and substances
* Having received radiotherapy and / or chemotherapy before surgery
* Having the disease that requires infective endocarditis prophylaxis (Rheumatic valve diseases, prosthetic heart valves, previous endocarditis, etc.)
* Corruption of cranium integrity and emergency surgery planned
* Having systemic or intracranial infections
* Transfenoidal surgery intervention planned
* Using implants during surgical intervention
* Using external ventricular drainage / lumbar drainage during and after surgical intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-10-03 (Estimated); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rate | Postoperative 90 days
  Within the postoperative 90 days, if there is purulent exudate or nonpurulent but culture was pozitive, we accepted them as Surgical Site Infection (SSI) diagnosed.
  Patient's case doctor will be responsible to document in date collection form, if there are surgical site infection occur. A research team is responsible for the data collection. The definition of surgical site infection will be according to CDC definitions of nosocomial surgical site infections: a modification of CDC definitions of surgical wound infection.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Özbaş, Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Department of Neurosurgery, Bakirkoy Research and Training Hospital for Neurology, Neurosurgery, and Psychiatry, İstanbul, Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided